CLINICAL TRIAL: NCT02105675
Title: Randomized, Open-label, Parallel-group, Multi-centre Phase II Clinical Trial of Active Cellular Immunotherapy With Preparation DCVAC/PCa in Patients With Castrate-resistant Prostate Cancer
Brief Title: Phase II Study of DCVAC/PCa Added to Standard Chemotherapy for Men With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP001; 2011-004735-32 (EudraCT Number)
Record Dates: First submitted 2014-03-24; First posted 2014-04-07 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2015-06

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic
Keywords: Immunotherapy; Metastatic; Castrate Resistant; Prostate Cancer; Biological; Vaccine
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCVAC/PCa add on to Standard of Care (Experimental): Combination therapy with Dendritic Cells DCVAC/PCa and Standard of Care
  Interventions: Biological: Dendritic Cells DCVAC/PCa
- Standard of Care (Active Comparator): Docetaxel as an Active Comparator
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Dendritic Cells DCVAC/PCa — DCVAC/PCa is the experimental therapy added on to Docetaxel
  Arms: DCVAC/PCa add on to Standard of Care
Drug: Docetaxel — Docetaxel is Standard of Care First Line Chemotherapy
  Other Names: taxotere
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine whether DCVAC/PCa added onto Standard of Care therapy can improve survival times for patients with Metastatic Castration Resistant Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥ 18 years
* Histologically confirmed prostate cancer
* Presence of skeletal metastasis (by CT or PET or MRI)
* Disease progression documented by increasing PSA or two new lesions
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2

Exclusion Criteria:

* Confirmed brain and/or leptomeningeal metastases
* Prior chemotherapy for prostate cancer
* Peripheral neuropathy of Common Toxicity Criteria (CTC) grade 2 or greater
* Other uncontrolled intercurrent illness
* Treatment with immunotherapy against PCa
* Clinically significant cardiovascular disease
* Active autoimmune disease requiring treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Survival rate | 135 weeks

SECONDARY OUTCOMES:
Radiographic Progression Free Survival | 135 weeks
Duration to Prostate Specific Antigen (PSA) Progression | 135 weeks
Changes in Quality of Life (QOL) assessed by European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 | 0, 10, 22, 37, 53, 65 weeks
Changes in Pain assessed by EORTC QLQ-C30 | 0, 10, 22, 37, 53, 65 weeks
Incidence of Adverse Events | 135 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Scheiner, PhD, Study Director — Sotio Biotech Inc.
Locations (10):
- Czechia (10):
  - Brno
  - Hradec Králové
  - Jihlava
  - Liberec
  - Nová Ves pod Pleší
  - Olomouc
  - Ostrava
  - Prague
  - Ústí nad Labem
  - Zlín

IPD SHARING:
Plan to Share IPD: Undecided
possibly shared on EMA website